CLINICAL TRIAL: NCT07158957
Title: WOMENinMOTION An Intervention Model for Pelvic Girdle Pain to Acquire Health-promoting Habits in Pregnancy and Prevent Chronic Pain in Women
Brief Title: WOMENinMOTION An Intervention Model for Pelvic Girdle Pain
Acronym: WIMPGP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Västra Götaland_WIMPGP; 2022-00146 (Other Grant/Funding Number: FORTE); VGRINN-979977 (Other Grant/Funding Number: Västra Götalandsregionens Innovationsfond); VGRINN-993309 (Other Grant/Funding Number: Västra Götalandsregionens Innovationsfond)
Record Dates: First submitted 2025-03-28; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2024-10

CONDITIONS: Pelvic Girdle Pain; Physical Activity
Keywords: pregnancy-related pelvic girdle pain; prevention of chronic pain; health-promotion; pain education; digital intervention,
MeSH Terms: conditions — Pelvic Girdle Pain; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- usual maternity health care + digital care (+when needed-WIM at physiotherapy clinic)) (Experimental): pregnant women who in addition to usual care get our model WOMENinMOTION (WIM) on a digital platform. When needed, referred to physiotherapy at clinic for WIM
  Interventions: Other: knowledge; Behavioral: motivation for behavioral change
- usual maternity health care (No Intervention): usual maternity health care according to regional guidelines including general advice

INTERVENTIONS:
Other: knowledge — -knowledge on pain in general and specifically pelvic girdle pain Pregnant women who in addition to usual care get our model WOMENinMOTION on a digital platform with self-directed content areas modules and linked tasks to promote physical activity and function by reducing concerns, pain, and building confidence for physical activity and realistic expectations.
  When women consider the digital platform insufficient, they are referred to physiotherapy at clinic for physiotherapeutically individually coached content of WIM
  Other Names: individual clinical physiotherapy
  Arms: usual maternity health care + digital care (+when needed-WIM at physiotherapy clinic))
Behavioral: motivation for behavioral change — motivation to be physically active
  Arms: usual maternity health care + digital care (+when needed-WIM at physiotherapy clinic))

SUMMARY:
The overall aim is to educate women to handle common pregnancy-related pain experiences to facilitate healthy life-long physical activity habits and prevent chronic pain.

Our developed WOMENinMOTION model with person-centred preventions and interventions focused on management of pain components added to usual care, will be evaluated in a randomized control study against usual care.

Data and method The model WOMENinMOTION is built on pain education and management of the sensory, emotional, and cognitive components of pain. Through pain management and motivation, pregnant women are guided to choose personal tools for health-promoting physical activity and adaptation of daily activities. Instructive films of exercises, pelvic belt application, and knowledge to meet worries are provided digitally. When the digital content is insufficient, the model is supported by physiotherapist.

Plan for project realisation WOMENinMOTION developed in collaboration with women with PGP, will be pilot tested including analysis of focus groups interviews 2024. The model is evaluated by self-reported questionnaires in a multicenter randomised controlled trial 2025-27 with primary outcomes: physical activity, function and health in gestational week 35, 4 months, 1 and 2 years after birth. Secondary outcomes is PGP prevalence, satisfaction with care, and health economy.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with or without pelvic girdle pain

Exclusion Criteria:

* previous fracture, malignancy or surgical interventions (pelvic floor, spine, pelvis, or hip) or disease of musculoskeletal-or nervous system
* serious intercurrent diseases such as diabetes and high blood pressure.
* multiple pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 592 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical activity: the Pregnancy Physical Activity Questionnaire | From enrollment to gestational weeks 35, 4 months, 1 and 3.5 years after birth
  different domains of physical activity in every day life
Health by EQ5D | From enrollment to gestational weeks 35, 4 months, 1 and 3.5 years after birth
  Health-related quality of life by the EuroQol 5-dimension questionnaire.
Function, summary of sensory components of pain | From enrollment to gestational weeks 35, 4 months, 1 and 3.5 years after birth
  SENSORY component of pain: Severity and disability of Pelvic Girdle Pain - measured by the Pelvic Girdle Questionnaire (PGQ).
Function, summary of cognitive components of pain | From enrollment to gestational weeks 35, 4 months, 1 and 3.5 years after birth
  COGNITIVE component of pain: Self-efficacy for carrying out physical activity - measured by the Pregnancy-Exercise Self-Efficacy Scale (P-ESES).
Function, summary of emotional components of pain | From enrollment to gestational weeks 35, 4 months, 1 and 3.5 years after birth
  EMOTIONAL component of pain: Concern about pain - a Numeric Rating Scale of 0-10.

SECONDARY OUTCOMES:
Person-centered function | From enrollment to gestational weeks 35, 4 months, 1 and 3.5 years after birth
  Person-centered function, assessed by the Patients Specific Function Scale (PSFS). Two, by the participant, self-chosen activities rated on a numeric rating scale of 0-10; 10 = have full function
Prevalence of pelvic girdle pain | From enrollment to gestational weeks 35, 4 months, 1 and 3.5 years after birth
  Prevalence of Pelvic Girdle Pain measured with self-administered pelvic pain provocation tests.
Work ability | From enrollment to gestational weeks 35, 4 months, 1 and 3.5 years after birth
  Work ability, measured by one question from the Work Ability Index.
Evening pain | From enrollment to gestational weeks 35, 4 months, 1 and 3.5 years after birth
  Evening pain intensity at its worst, measured by a NRS where 10 = worst pain
Pain frequency | From enrollment to gestational weeks 35, 4 months, 1 and 3.5 years after birth
  Pain frequency by question
Depressive symptoms | From enrollment to gestational weeks 35, 4 months, 1 and 3.5 years after birth
  Symptoms of depression, measured by the Edinburgh Postnatal Depression Scale
health economy | From enrollment to gestational weeks 35, 4 months, 1 and 3.5 years after birth
  Health-economy evaluation with direct/indirect costs (days on sick leave, visits to health care providers).

OTHER OUTCOMES:
Fear avoidance belief | From enrollment to gestational weeks 35, 4 months, 1 and 3.5 years after birth
  Fear avoidance beliefs questionnaire subscale that measures physical activity (FABQ-PA). Zero is equivalent to no fear avoidance and 24 indicates the highest possible fear avoidance.
Catastrophizing thoughts | From enrollment to gestational weeks 35, 4 months, 1 and 3.5 years after birth
  Using- Pain Catastrophizing Scale, ranging from 0 (never) to 4 (always). The total score is the sum of the scores for the individual items, and ranges from 0 (no catastrophizing thoughts) to 52 (highest possible catastrophizing thoughts)

CONTACTS AND LOCATIONS:
Overall Officials: Annelie Gutke, PhD, associate professor, Principal Investigator — Göteborg University
Locations (2):
- Sweden (2):
  - Närhälsan Gibraltargatan rehabmottagning, Gothenburg
  - Närhälsan Eriksberg rehabmottagning, Gothenburg

IPD SHARING:
Plan to Share IPD: No